CLINICAL TRIAL: NCT07281963
Title: Chilipad Sleep Optimization Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Efforia, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 13228
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Single Arm observational where participants act as their own control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Single arm where participants act as their own control (Experimental): Single arm where participants act as their own control
  Interventions: Device: Chilipad Dock Pro Bed Cooling System and Sleep Tracker

INTERVENTIONS:
Device: Chilipad Dock Pro Bed Cooling System and Sleep Tracker — The Chilipad Dock Pro Bundle is an advanced sleep system designed to optimize sleep by dynamically adjusting the bed's surface temperature. It consists of a thermoregulated mattress pad and a Dock Pro control unit that actively circulates water through the pad, allowing users to customize the temperature between 55°F and 115°F. The system offers both single and dual control, making it ideal for individual or shared use. Equipped with AI-driven features, the Dock Pro can monitor sleep patterns and environmental factors to make real-time adjustments, ensuring optimal sleep conditions throughout the night. This intelligent temperature management system is only enhanced when paired with the optional Sleepme Tracker, creating a personalized sleep experience.

SUMMARY:
This study evaluates the Chilipad Dock Pro Bed Cooling System and Sleep Tracker, examining how bed temperature influences sleep quality and overall well-being.

DETAILED DESCRIPTION:
This remotely administered decentralized trial is designed to rigorously evaluate the impact of the Chilipad Dock Pro Bed Cooling System on sleep quality and overall well-being. In a world where optimal sleep remains elusive for many, this study seeks to provide evidence-based insights into how temperature regulation can significantly affect restful nights. Leveraging the potential of the Chilipad Dock Pro Bed Cooling System, which offers personalized temperature settings aimed at enhancing the sleep environment, this research focuses on quantifying its effectiveness through scientifically validated metrics.

Participants in this study will engage in a comprehensive assessment process, utilizing the PROMIS Sleep Disturbance Scale, Well-being Survey, and SF-36 as primary tools for measuring outcomes. By collecting data remotely from participants in their natural sleep settings, this trial aims to offer a real-world evaluation of the system's capability to improve sleep quality. From baseline to endpoint, the study will monitor changes in sleep disturbance, overall well-being, and health-related quality of life, providing a robust dataset for analysis.

The overarching objective of this research is to empower participants with concrete, science-backed data on the impact of the Chilipad Dock Pro Bed Cooling System on their sleep and well-being. By the conclusion of the study, participants will have access to measurable insights into how the system has influenced their sleep patterns and quality of life, thereby aiding in informed decision-making for enhanced health outcomes.

Furthermore, this study stands to significantly contribute to the broader scientific and healthcare communities by establishing a clear link between temperature regulation during sleep and sleep quality improvements. In addressing the gap between anecdotal evidence and scientific validation, the findings from this research are anticipated to underscore the importance of sleep environment optimization. By demonstrating the efficacy of the Chilipad Dock Pro Bed Cooling System through significant changes in validated measures of sleep and well-being, this study could pave the way for revolutionary approaches in sleep health management, acknowledging the limitations posed by individual sleep needs variability and external environmental factors.

ELIGIBILITY:
Inclusion Criteria:

* Can read and understand English.
* US resident.
* Willing and able to follow the requirements of the protocol.

Exclusion Criteria:

* Individuals with concerns about water leakage.
* Individuals with sleep disorders related to changes in temperature
* Individuals with thermal sensitivity
* Individuals who are easily frustrated by technology.
* Individuals with pacemakers or medical implants sensitive to electromagnetic fields
* Pregnant individuals

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-09-25 (Estimated); Study Completion 2026-09-25 (Estimated)

PRIMARY OUTCOMES:
PROMIS Sleep Disturbance Scale | Change from baseline (Day 1-3) in PROMIS Sleep Disturbance Scale at 4 weeks after the start of the intervention (Day 27-33)
  The PROMIS Sleep Disturbance Scale is a validated and widely used assessment tool developed as part of the Patient-Reported Outcomes Measurement Information System (PROMIS) initiative. It is designed to measure the severity of sleep disturbances and disruptions experienced by individuals. This scale includes a range of questions that assess the frequency and impact of various sleep-related issues, such as difficulty falling asleep, nighttime awakenings, and restless sleep. Healthcare professionals and researchers rely on this scale to better understand and quantify sleep problems in patients, enabling them to tailor interventions and treatment strategies to address sleep-related concerns effectively.
Well-being Survey | Change from baseline (Day 1-3) in Well-being Survey at 4 weeks after the start of the intervention (Day 27-33)
  Please answer the following questions to assess your well-being.
36-Item Short Form Survey Instrument (SF-36) | Change from baseline (Day 1) in SF-36 at 4 weeks after the start of the intervention (Day 29-31)
  The SF-36, or Short Form 36, is a widely used health-related quality of life questionnaire that consists of 36 questions designed to assess a person's physical and mental well-being. It measures various aspects of an individual's health, including physical functioning, role limitations due to physical and emotional problems, social functioning, mental health, energy and vitality, pain, and general health perceptions. The SF-36 provides a comprehensive overview of a person's health status and is frequently used in clinical research, healthcare assessments, and population health studies. Its versatility and ability to assess multiple dimensions of health make it a valuable tool for evaluating the impact of medical interventions and health-related interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- Efforia, New York, New York, United States

REFERENCES:
- See also: Additional information and join instructions on Efforia — https://app.efforia.com/wp-admin/admin.php?page=llms-course-builder&course_id=13223